CLINICAL TRIAL: NCT06172140
Title: Efficacy and Safety of Ciprofol for the Sedation in Patients Undergoing Hysteroscopy: A Prospective, Randomized, Non-inferiority Trial.
Brief Title: Efficacy and Safety of Ciprofol for the Sedation in Patients Undergoing Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2023-1091-02
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Ciprofol; Hysteroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol group (Experimental): Intravenous injection of ciprofol
  Interventions: Drug: Ciprofol group
- Propofol group (Experimental): Intravenous injection of propofol
  Interventions: Drug: Propofol group

INTERVENTIONS:
Drug: Ciprofol group — All patients received 5 μ g of sufentanil 1 minute before intravenous infusion of ciprofol, followed by intravenous injection of ciprofol (0.4mg/kg). When the MOAA/S score is ≤ 1, vaginal disinfection begins. During the induction of sedation, the MOAA/S score is evaluated every 30 seconds. If the MOAA/S score remains above 1, a supplementary dose of 1/2 of the initial dose is injected within 10 seconds. During the maintenance phase, supplementary doses are given when there are signs of physical activity, eye opening, or speech. If more than 5 additional doses are required within 15 minutes, painless hysteroscopy is considered a failure, and propofol is immediately used to enhance sedation.
  Arms: Ciprofol group
Drug: Propofol group — All patients received 5 μ g of sufentanil 1 minute before intravenous infusion of propofol, followed by intravenous injection of propofol (2 mg/kg) for 30 seconds. When the MOAA/S score is ≤ 1, vaginal disinfection begins. During the induction of sedation, the MOAA/S score is evaluated every 30 seconds. If the MOAA/S score remains above 1, a supplementary dose of 1/2 of the initial dose is injected within 10 seconds. During the maintenance phase, supplementary doses are given when there are signs of physical activity, eye opening, or speech. If more than 5 additional doses are required within 15 minutes, painless hysteroscopy is considered a failure, and propofol is immediately used to enhance sedation.
  Arms: Propofol group

SUMMARY:
Eligible patients undergoing hysteroscopy were randomly assigned in a 1:1 ratio to receive intravenous anesthesia with either propofol (2 mg/kg) or remifentanil (0.4 mg/kg).Continuous monitoring of pulse oximetry (SpO2), blood pressure (BP), heart rate (HR), expired gas partial pressure of carbon dioxide, integrated respiratory index (IPI), tidal volume (TV), respiratory rate (RR), and minute ventilation (MV) was performed.During induction, the MOAA/S score was assessed every 30 seconds. If the MOAA/S score remained >1, a supplementary dose of 1/2 of the initial dose was injected within 10 seconds.If more than 5 supplementary doses were required within 15 minutes, it was considered that the painless hysteroscopy failed and propofol was used to enhance sedation.Continuous oxygen administration at a flow rate of 5 liters per minute was provided through nasal catheters until the patient was fully alert with a MOAA/S score of 5 and vital signs were stable.Observation indicators included: (1) the success rate of hysteroscopy;(2) induction time (MOAA/S ≤ 1 after the first dose);(3) full recovery time of consciousness;(4) operation duration;(5) number of additional anesthetics;(6) incidence of hypotension, hypoxemia, sinus bradycardia, delayed recovery, and injection pain;(7) respiratory parameters and minimum SpO2, IPI values before anesthesia, after induction, and after awakening.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent form
* Stable vital signs and qualified anesthesia outpatient evaluation
* No contraindications to anesthesia

Exclusion Criteria:

* Not willing to sign informed consent form
* Anaesthesia drug allergy
* Severe central nervous system diseases
* Severe hypertension and diabetes
* Mental disorders
* History of using psychotropic drugs in the past 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Success rate of painless hysteroscopy | During procedure (The inspection is completed and the vaginal speculum is removed)
  During the induction of sedation, the anaesthesiologist evaluated the MOAA/S score every 30 s. If the MOAA/S score remained >1 after 2 min of initial administration of the study drug, a top-up dose of 1/2 the initial dose was injected over 10 s. During the maintenance phase, supplementary doses are given when the MOAA/S score is>1, and repeated every 2 minutes as needed. If more than 5 additional doses are required within 15 minutes, it is considered a failure of painless hysteroscopy .

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Sun Yat-sen Memorial Hospital, Sun Yat-sen Universit, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng S, Wu H, Liu Z, Liu D, Cao M, Fu G. Efficacy and safety of ciprofol for sedation/anesthesia in patients undergoing hysteroscopy: a prospective, randomized, non-inferiority trial. Ann Med. 2025 Dec;57(1):2517820. doi: 10.1080/07853890.2025.2517820. Epub 2025 Jun 18. PMID 40530830